CLINICAL TRIAL: NCT02904421
Title: A Six Years Longitudinal Cohort Study on the Changes in Bone Density, Bone Quality and Its Association With Bone Turnover Markers and Curve Severity in Adolescent Idiopathic Scoliosis With and Without 2 Years of Calcium and Vit-D Supplementation
Brief Title: 6 Years Study on Changes in Bone Quality, Bone Turnover and Curve Severity in AIS With and Without Calcium and Vit-D Supplementation
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz-ping Lam, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CALTC4_v1
Record Dates: First submitted 2016-09-04; First posted 2016-09-19 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Scoliosis; Vitamin D; Bone
Keywords: scoliosis; spinal deformity; vitamin D; bone health
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: the placebo group
- Group 2: the low-dose treatment group with 600mg calcium + 400IU Vit-D3/day
- Group 3: the high-dose treatment group with 600mg calcium + 800IU Vit-D3/day

SUMMARY:
The study aimed to:

1. To investigate and compare the changes in bone mineral density (BMD), trabecular bone micro-architecture, bone strength, and curve severity at a mean of 6 years longitudinal follow up in AIS girls with low bone mass between Group A and B:

   1. Group A: subjects followed at a mean of 4 years after completion of 2-year calcium and Vit-D supplementation and
   2. Group B: subjects without calcium and Vit-D supplementation
2. To evaluate the correlation between changes in BMD, trabecular bone micro-architecture, and bone strength documented in Objective 1 with changes in serum bone turnover markers

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a complex three-dimensional spinal deformity mostly affecting girls in the peri-pubertal period. Prevalence ranges from 2 to 4% in the general population. When the deformity becomes severe, serious morbidities can occur including early back degeneration, cardiopulmonary compromise, grossly deformed torso and associated psychosocial issues which could pose serious health threats for these young patients.

One important health threat that deserves special attention is osteopenia as defined by Bowden et al. for children having BMD age and gender-adjusted Z-score < -1. 30-38% of AIS girls were osteopenic. Osteopenia could persist across puberty and was found to be a significant and independent prognostic factor for curve progression in AIS. Osteopenia was also found to be associated with low dietary calcium (Ca) intake at a median of 400mg/day among AIS girls. The low Ca intake was significantly correlated with age-adjusted peripheral volumetric bone mineral density (vBMD) measured by peripheral quantitative computed tomography (pQCT), as well as axial and peripheral areal BMD (aBMD) measured by Dual-Energy X-ray Absorptiometry (DXA).

Low calcium intake when coupled with low Vit-D status can seriously affect a child's bone health. Without Vit-D, only 10 to 15% of dietary calcium is absorbed, and 1,25-(OH)2Vit-D can increase intestinal calcium absorption to 30-40%. Vit-D insufficiency or disturbance in Vit-D physiology is associated with osteopenia, deranged muscle function and ligamentous laxity which could potentially predispose AIS subjects to curve progression.

Given that serum 25(OH)Vit-D level was also found to be low at a mean level of 41.6 nmol/L among AIS subjects, our group has conducted the first 2-year randomized double-blinded placebo-controlled trial using calcium and Vit-D supplementation for young AIS girls with low bone mass (the Cal study). There were three study groups in the trial, namely Group 1 (the placebo group), Group 2 (the low-dose treatment group with 600mg calcium + 400IU Vit-D3/day) and Group 3 (the high-dose treatment group with 600mg calcium + 800IU Vit-D3/day). The study showed strong evidences of positive bone accretion effects and therapeutic control of curve progression in groups with supplementation (Group 2 and 3). Following the therapeutic gain in BMD and improvement in bone quality with 2-year intervention with calcium and Vit-D supplementation, it will be important to evaluate if the effects persist after supplement withdrawal. This study would help to address this key issue by evaluating whether the beneficial effects of 2-year calcium and Vit-D supplementation persist at an average of 4 years after withdrawal of supplementation. The BMD, trabecular bone micro-architecture, bone strength, image-based and serum bone turnover parameters, and curve severity at 4 years after withdrawal of supplement would be compared with measurements done before and at end of supplementation.

Outcome of this study will provide important scientific data on the long term effects of 2-year calcium and Vit-D supplementation, thus justifying the need of lifestyle modification, duration and dose of supplementation for better bone health and curve control in adolescents suffering from AIS. If the beneficial effects are proven to be sustainable, the 2-year calcium and Vit-D supplements can be incorporated into the treatment protocol for AIS not only in Hong Kong, but also in Mainland China and other parts of the world; otherwise longer period of supplementation for sustained positive bone accretion effects and prevention of curve progression will be desirable for attaining peak bone mass and curve control to prevent osteopenia-related and scoliosis-related complications when approaching adulthood.

This six years longitudinal follow-up study with 2-year active supplementation period and 4-year post-withdrawal follow up for this cohort of adolescent girls is unique. Not only are the effects of calcium and vitamin D supplementation being followed, the placebo group in the original clinical trial provides the longitudinal changes on anthropometric, bone density, bone quality parameters and curve severity which will yield important reference information for local adolescents with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from the Cal study

Exclusion Criteria:

* Subjects that are pregnant
* Subjects with fracture

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All 330 subjects from the Cal study will be invited to participate. Order of recruitment will follow the order of recruitment during the initial study at a first-entry first-serve basis.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2016-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline clinical features of scoliosis at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  A long standard standing postero-anterior (PA) whole spine radiograph will be used for grading curve severity in terms of Cobb angle according to the standard Cobb method.
Change from baseline BMD Measurement at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  Areal BMD (g/cm2) and BMC (g/cm) of bilateral hips (femoral neck) will be measured by DXA.
Change from baseline volumetric BMD (vBMD), bone geometry and trabecular bone micro-architecture at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  Detailed bone measurement of the non-dominant distal radius will be carried out with the in-vivo HR-pQCT using an established measurement protocol.
Change from baseline bone mechanical strength at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  Finite element analysis (FEA) will be used to assess the bone strength non-invasively. Finite element (FE) models of the radius will be created directly from the HR-pQCT images using Scanco FE solver integrated in the IPL software.
Change from baseline biochemical markers for bone formation and resorption at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  Serum P1NP and β-CTx will be assayed to determine bone formation and resorption activity.
Change from baseline serum Vitamin D concentration at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  Serum 25(OH)Vit-D concentrations will be measured by liquid chromatography isotope-dilution electrospray ionization tandem mass spectrometry (LCTMS).

SECONDARY OUTCOMES:
Change from baseline dietary intakes and physical activity at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  The dietary intake and physical activity data are recorded as covariates for statistical analysis on bone changes of the study groups.
Change from baseline anthropometric measurements and maturity assessment at end of 2 year supplementation and at 4 years post-treatment follow up | baseline, end of 2 year supplementation, 4 years post-treatment follow up
  Detail anthropometric measurements including body height, weight, arm span will be measured with standard stadiometry techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ping Lam, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology, Prince of Wales Hospital, Hong Kong, Hong Kong, China